CLINICAL TRIAL: NCT07136376
Title: B-challenged: A Multi-actor Approach in Creating Safe and Attractive Physical and Social Environments to Promote Children's Active Outdoor Play and Healthy Dietary Behaviours
Brief Title: B-challenged: Co-creating Physical and Social Environments to Promote Children's Active Outdoor Play
Acronym: B-challenged
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: University of Southern Denmark, Odense, Denmark (Unknown); Fundación Instituto Investigación Sanitaria Aragón, Zaragoza, Spain (Unknown); Institute of Mother and Child, Warshaw, Poland (Unknown); University of Bremen, Leibniz Institute for Prevention Research and Epidemiology, Bremen, Germany (Unknown); Foundation of the Institute of Mother and Child, Warsaw, Poland (Unknown)
Responsible Party: Principal Investigator, Teatske Altenburg, A/Prof., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: "HEALTHEQUITY-039 B-challenged
Record Dates: First submitted 2025-07-02; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Active Outdoor Play and Related Healthy Dietary Behaviours
Keywords: Participatory Action Research; System dynamics; Child co-researcher; Lifestyle behaviours; Multi-actor collaborations
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children growing up in underserved neighbourhoods. (Experimental)
  Interventions: Other: Physical and social environmental interventions.

INTERVENTIONS:
Other: Physical and social environmental interventions. — To be determined in the co-creation groups at the five sites (Denmark, Germany, Poland, Spain, the Netherlands)

SUMMARY:
BACKGROUND An alarmingly low number of children meet public health guidelines for physical activity and healthy dietary behaviours, and are at increased risk of developing lifestyle-related diseases. Importantly, this burden is already unequally distributed at an early age. Unhealthy lifestyle behaviours are driven by complex mechanisms that differ across boys and girls growing up under different socio-economic circumstances. Outdoor play is an important contributor to children's levels of physical activity. Yet, children growing up in underprivileged neighbourhoods play less outside due to limited access to safe and attractive outdoor spaces and appropriate and affordable after school activities than other children. At the same time, today's children have abundant access to inexpensive energy-dense foods and online sedentary activities.

AIM B-challenged aims to tackle the complexity of equality in children's active outdoor play and healthy dietary behaviours by co-creating, implementing and evaluating interventions in the physical and social environmental together with children growing up in socio-economically underprivileged neighbourhoods and other key actors.

APPROACH B-challenged introduces a multi-actor, inter-sectorial democratic approach in five European countries (Denmark, Germany, Spain, Poland and the Netherlands), including all key actors (e.g. children, parents, teachers, policy makers). The investigators in B-Challenged will closely collaborate with all key actors, conduct analyses in European cohort data and consider the broader system (e.g. neighbourhood, family) as well as previous lessons-learned. Therewith, B-challenged aims at structural, relevant and feasible improvements in the physical and social environment promoting children's active outdoor play and dietary behaviours. B-challenged will impact all key actors in the selected neighbourhoods and far beyond through disseminating protocols and recommendations (research and policy) for upscaling the B-challenged approach.

ELIGIBILITY:
Inclusion criteria child co-researchers:

* Living in a underserved urban neighbourhood
* Aged 9-12 years

Inclusion criteria children participating in the effect evaluation:

* Living in the same underserved neighbourhood as the child co-researchers
* Aged 6-12 years

Inclusion criteria adult actors:

* Based on results of the actor mapping (including adult actors interview 1 and adult actors recruitment form)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Time spent in outdoor play | Baseline and 12 months follow up (i.e., after intervention implementation).
  Time spent in outdoor play is assessed by a child-questionnaire (based on HBSC questionnaire, US national Kids Survey, and nationwide survey from Norway) and covers active travel, organised outdoor activities and unorganised outdoor play.
  Duration reported using 6 response options (longer duration of outdoor play contributing to a healthier lifestyle): 0-½ hour; ½-1 hour; 1-1 ½ hour; 1 ½-2 hours; and More than 2 hours.

SECONDARY OUTCOMES:
Frequency of fruit consumption during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire item on the frequency of consumption of fruits during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of fruit consumption contributes to a healthy lifestyle.
Frequency of vegetable consumption during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire item on the frequency of consumption of vegetables during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of vegetable consumption contributes to a healthy lifestyle.
Frequency of consumption of sweets during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire item on the frequency of consumption of sweets (candy or chocolate) during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of consumption of sweets contributes to a more unhealthy lifestyle.
Frequency of consumption of crisps and other salty snacks during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire items on the frequency of consumption of crisps and other salty snacks during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of crisps and other salty snacks consumption contributes to a more unhealthy lifestyle.
Frequency of consumption of coke or other soft drinks that contain sugar during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire items on the frequency of consumption of coke or other soft drinks that contain sugar during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of consumption of coke or other soft drinks that contain sugar contributes to a more unhealthy lifestyle.
Frequency of consumption of fast-food (pizza, kebab, burgers) during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire items on the frequency of consumption of fast-food (pizza, kebab, burgers) during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of fast-food (pizza, kebab, burgers) consumption contributes to a more unhealthy lifestyle.
Frequency of consumption of energy drinks (such as Red Bull) during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire items on the frequency of consumption of energy drinks (such as Red Bull) during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of energy drinks (such as Red Bull) consumption contributes to a more unhealthy lifestyle.
Frequency of consumption of water during outdoor play, assessed by: | Baseline and 12 months follow up (i.e., after intervention implementation)
  Child-questionnaire items on the frequency of consumption of water during outdoor play, partially based on the HBSC questionnaire, the US national Kids Survey and a nationwide survey from Norway.
  Frequency reported on a 7-point scale: Never Less than once a week; Once a week; 2-4 days a week; 5-6 days a week; Once a day, every day; Every day, more than once.
  Higher frequency of water consumption contributes to a healthy lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Teatske Altenburg, A/Prof, Principal Investigator — Amsterdam UMC, location VUmc, Amsterdam, the Netherlands
Locations (5):
- University of Southern Denmark, Odense, Denmark
- University of Bremen, Leibniz Institute for Prevention Research and Epidemiology, Bremen, Germany
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands
- Institute of Mother and Child, Warsaw, Poland
- Fundación Instituto Investigación Sanitaria Aragón, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
B-Challenged uses the approach "as open as possible, as restricted as necessary" as the leading principle in providing open access to research data, which includes taking measures to make research data findable, accessible, interoperable and reusable.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting from June 2025.
Access Criteria: Only anonimized data will be shared as well as additional supporting information, such as a co-creation protocol, data dictionary code book, topic lists for focus groups and interviews, etc.
URL: https://osf.io/nd6ky/